CLINICAL TRIAL: NCT05137314
Title: A Phase 1b Open-Label, Dose-Escalating Study to Evaluate the Safety and Tolerability of PLG0206 in Patients Undergoing Debridement, Antibiotics, and Implant Retention (DAIR) for Treatment of a Periprosthetic Joint Infection (PJI) Occurring After Total Knee Arthroplasty (TKA)
Brief Title: Study in Patients Undergoing Debridement, Antibiotics, and Implant Retention (DAIR) for Treatment of a Periprosthetic Joint Infection (PJI) Occurring After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptilogics (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLG0206-PJI-101
Record Dates: First submitted 2021-10-28; First posted 2021-11-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Joint Infection
Keywords: PJI; knee infection

STUDY DESIGN:
Intervention Model Description: Open-Label, Dose-Escalating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3 mg/mL PLG0206 (Experimental): administered intraoperatively by local irrigation
  Interventions: Drug: PLG0206
- 10 mg/mL PLG0206 (Experimental): administered intraoperatively by local irrigation
  Interventions: Drug: PLG0206

INTERVENTIONS:
Drug: PLG0206 — PLG0206 is an engineered antibacterial peptide (EAP)

SUMMARY:
The purpose of this study is to learn about the safety and effects of PLG0206 for treating periprosthetic joint infections (PJI) in conjunction with the DAIR (debridement, antibiotics and implant retention) surgical procedure for patients with periprosthetic joint infections (PJI) after total knee arthroplasty (TKA) .

DETAILED DESCRIPTION:
Peptilogics, Inc. is developing PLG0206 for the treatment of PJIs. PLG0206 is an engineered antibacterial peptide (EAP) based on naturally-occurring antimicrobial peptides (AMPs). Recent work on PLG0206 has documented that PLG0206 is a highly effective anti-biofilm agent, in addition to its established activity against planktonic staphylococcus, both in vitro and in a murine animal model of PJI.

PLG0206 will be investigated in this study for treatment of PJI in conjunction with the DAIR procedure followed by the 6-week course of antimicrobial therapy that is standard-of-care (SOC) in this indication.

Patients will be followed for approximately 1 year post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-fixed prosthesis;
* Patients who have a pre- or intra-operative diagnosis of TKA-PJI

Exclusion Criteria:

* Patients for whom a DAIR procedure is not indicated;
* Patients with loose prosthesis and/or surgical treatment requiring removal of well-fixed, non-modular implants at screening;
* Patients with previous history or presence of osteomyelitis in the index limb;
* Patients who have uncontrolled diabetes mellitus;
* Patients with body mass index >50 kg/m2 at screening;
* Patients who are immunosuppressed;
* Patients who require therapeutic anticoagulation and/or antiplatelet therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
The percentage of treatment emergent AEs | approximately 1 year
  the safety and tolerability of PLG0206 administered via an irrigation solution for the treatment of a PJI occurring after TKA during DAIR.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Stanford Hospital, Palo Alto, California
  - Gulfcoast Research, Sarasota, Florida
  - LifeBridge, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - NYU Langone Orthopedic Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Rothman, Philadelphia, Pennsylvania
  - Memorial Hermann Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - WVU, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No